CLINICAL TRIAL: NCT06261801
Title: Efficacy of Electroacupuncture Combined With Pregabalin in the Treatment of Trigeminal Herpetic Neuralgia: a Multicenter Randomized Controlled Trial Study Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third People's Hospital of Hangzhou (Other)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Ling Pin, Chief physician, The Third People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZY-ZJ-KJ-23088
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Trigeminal Herpetic Neuralgia
Keywords: Electroacupuncture; pain; randomized controlled trial; protocol
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medication Group (Active Comparator): Participants in the medication group would take 150-mg pregabalin capsules orally twice daily (total daily dose, 300 mg) for 4 weeks. The follow-up period is 3 months.
  Interventions: Other: Medication Group
- EA Group (Experimental): The subjects in this group will receive 3 times per week, and 4 weeks of continuous intervention for a total of 12 times. The follow-up period is 3 months.
  Interventions: Other: EA Group
- EA+Medication Group (Experimental): The subjects in this group will receive 3 times per week, and 4 weeks of continuous intervention for a total of 12 times. The intervention including electroacupuncture(EA) treatment and combined with pregabalin (0.15g each time, twice daily). The follow-up period is 3 months.
  Interventions: Other: EA+Medication Group

INTERVENTIONS:
Other: Medication Group — Participants in the medication group would take 150-mg pregabalin capsules (manufactured by Pfizer Pharmaceuticals Co., Ltd) orally twice daily (total daily dose, 300 mg) for 4 weeks.
  Arms: Medication Group
Other: EA Group — Acupoints selection: Ashi acupoint, Sibai acupoint (ST2), Xiaguan acupoint (ST7), and Dicang acupoint (ST4) on the affected side. Acupoints for the diseased branches (all taken from the affected side): eye branch and Tongziliao point (GB1), the maxillary branch is taken from the Quanliao point (SI18), and the mandibular branch is taken from the Jiache point (ST6).Shenting point (DU24), Baihui point (DU20), Hegu point (LI4), Waiguan point (TE5), Yanglingquan point (GB34), and Taichong point (LR3) on the affected side Operation: The EA apparatus will be applied on the Ashi point and (LI4 - TE5). The treatment will last for 30 minutes and the electrical stimulation will be set as 2/100Hz in frequency.
  Arms: EA Group
Other: EA+Medication Group — Participants in the EA+Medication group would receive both EA and medical treatement. The acupoints and their location, needles, the settings of the EA device are the same as EA Group's; in the meanwhile, the medication and its dosage is the same as Medication Group's.
  Arms: EA+Medication Group

SUMMARY:
Trigeminal herpetic neuralgia is a common type of Zoster-associated Pain (ZAP), which troubles individuals in all ages and burdens society all over the world. Eleactroaupuncture (EA) is increasingly used in the treatment of ZAP due to its advantages such as low price, high safety, no adverse reactions, and high patient acceptance. Therefore, it is necessary to conduct randomized controlled trials to evaluate the effectiveness and safety of EA on ZAP and whether EA can be used as a substitute for pregabalin.

DETAILED DESCRIPTION:
Trigeminal herpetic neuralgia is a common type of Zoster-associated Pain (ZAP), which troubles individuals in all ages and burdens society all over the world. Eleactroaupuncture (EA) is increasingly used in the treatment of ZAP due to its advantages such as low price, high safety, no adverse reactions, and high patient acceptance. Therefore, it is necessary to conduct randomized controlled trials to evaluate the effectiveness and safety of EA on ZAP and whether EA can be used as a substitute for pregabalin.

ELIGIBILITY:
Inclusion Criteria:

1. meet the aforementioned diagnostic criteria for trigeminal ZAP, with a disease duration of 1 to 3 months;
2. have a visual analog scale (VAS) score of 4 points ≤ VAS ≤ 7 points;
3. be between 18 and 85 years old, regardless of gender;
4. have clear consciousness, the ability to distinguish pain, and complete basic communication;
5. voluntarily participate in the study, sign a written informed consent form, and fully understand the plan.

Exclusion Criteria:

1. do not meet the above-mentioned inclusion criteria;
2. have concomitant herpes zoster on the trunk or extremities, or other special types of herpes zoster like meningeal herpes zoster or visceral herpes zoster;
3. are pregnant or lactating patients;
4. are allergic to pregabalin or acupuncture stimulation;
5. have severe organ damage, cognitive dysfunction, mental disorder, aphasia, or other serious diseases that hinder cooperation with treatment;
6. have severe skin diseases;
7. have a pacemaker;
8. have been or are currently participating in other clinical studies within the past 3 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score change | Weeks 0 (baseline), Week 2 (Treatment), Week 4 (Treatment), Week 8 (Follow-up), and Week 16 (Follow-up)
  Intensity of pain range (lately 3 days' average): 0 =no pain to 10 =worst possible pain. Higher score indicating severe pain.

SECONDARY OUTCOMES:
McGill Pain Questionnaire Short Form (SF-MPQ) | Weeks 0 (baseline), Week 2 (Treatment), Week 4 (Treatment), Week 8 (Follow-up), and Week 16 (Follow-up)
  SF-MPQ focuses on the characteristics, intensity, syndrome and changes of pain during treatment without taking too much time, so it can sensitively reflect clinical changes and reflect the effectiveness of treatment.
Brief Pain Inventory Scale (BPI-SF) | Weeks 0 (baseline), Week 2 (Treatment), Week 4 (Treatment), Week 8 (Follow-up), and Week 16 (Follow-up)
  BPI-SF includes descriptive words such as the cause of pain, nature of pain, impact on life, and location of pain, which are used to describe the degree of pain and evaluate pain in various aspects.
Medical Outcomes Study Sleep Scale (MOS-SS) | Weeks 0 (baseline), Week 2 (Treatment), Week 4 (Treatment), Week 8 (Follow-up), and Week 16 (Follow-up)
  The MOS-SS consists of 12 items related to sleep quality over a 4-week recall period.
Hamilton Depression Rating Scale (HAMD)Hamilton Anxiety Rating Scale (HAMA) | Weeks 0 (baseline), Week 2 (Treatment), Week 4 (Treatment), Week 8 (Follow-up), and Week 16 (Follow-up)
  HAMA will be used to assess the anxiety status of the participants
Hamilton Depression Rating Scale (HAMD) | Weeks 0 (baseline), Week 2 (Treatment), Week 4 (Treatment), Week 8 (Follow-up), and Week 16 (Follow-up)
  HAMD will be used to assess the depression status of the participants
Short Form 36 Health Survey (SF-36) | Weeks 0 (baseline), Week 2 (Treatment), Week 4 (Treatment), Week 8 (Follow-up), and Week 16 (Follow-up)
  The SF-36 is a questionnaire with proven reliability and validity and is widely used to assess people's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Pin Lin, Study Director — The Hangzhou Third People's Hospital
Locations (1):
- The Hangzhou Third People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Werner RN, Nikkels AF, Marinovic B, Schafer M, Czarnecka-Operacz M, Agius AM, Bata-Csorgo Z, Breuer J, Girolomoni G, Gross GE, Langan S, Lapid-Gortzak R, Lesser TH, Pleyer U, Sellner J, Verjans GM, Wutzler P, Dressler C, Erdmann R, Rosumeck S, Nast A. European consensus-based (S2k) Guideline on the Management of Herpes Zoster - guided by the European Dermatology Forum (EDF) in cooperation with the European Academy of Dermatology and Venereology (EADV), Part 2: Treatment. J Eur Acad Dermatol Venereol. 2017 Jan;31(1):20-29. doi: 10.1111/jdv.13957. Epub 2016 Nov 2. PMID 27579792
- [Result] Johnson RW, Rice AS. Clinical practice. Postherpetic neuralgia. N Engl J Med. 2014 Oct 16;371(16):1526-33. doi: 10.1056/NEJMcp1403062. No abstract available. PMID 25317872
- [Result] Wood M. Understanding pain in herpes zoster: an essential for optimizing treatment. J Infect Dis. 2002 Oct 15;186 Suppl 1:S78-82. doi: 10.1086/342958. PMID 12353191
- [Result] Kawai K, Gebremeskel BG, Acosta CJ. Systematic review of incidence and complications of herpes zoster: towards a global perspective. BMJ Open. 2014 Jun 10;4(6):e004833. doi: 10.1136/bmjopen-2014-004833. PMID 24916088
- [Result] Gan EY, Tian EA, Tey HL. Management of herpes zoster and post-herpetic neuralgia. Am J Clin Dermatol. 2013 Apr;14(2):77-85. doi: 10.1007/s40257-013-0011-2. PMID 23456596
- [Result] Oster G, Harding G, Dukes E, Edelsberg J, Cleary PD. Pain, medication use, and health-related quality of life in older persons with postherpetic neuralgia: results from a population-based survey. J Pain. 2005 Jun;6(6):356-63. doi: 10.1016/j.jpain.2005.01.359. PMID 15943957
- [Result] Dubinsky RM, Kabbani H, El-Chami Z, Boutwell C, Ali H; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter: treatment of postherpetic neuralgia: an evidence-based report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2004 Sep 28;63(6):959-65. doi: 10.1212/01.wnl.0000140708.62856.72. PMID 15452284
- [Result] Dworkin RH, O'Connor AB, Kent J, Mackey SC, Raja SN, Stacey BR, Levy RM, Backonja M, Baron R, Harke H, Loeser JD, Treede RD, Turk DC, Wells CD. Interventional management of neuropathic pain: NeuPSIG recommendations. Pain. 2013 Nov;154(11):2249-2261. doi: 10.1016/j.pain.2013.06.004. Epub 2013 Jun 6. PMID 23748119